CLINICAL TRIAL: NCT01727557
Title: Anesthetic Technique for AV Fistulae Creation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accural Rate
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Naum Shaparin, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-08-302
Record Dates: First submitted 2012-06-08; First posted 2012-11-16 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Hemodialysis and AV fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Anesthesia, Conduction; Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anesthesia (Active Comparator)
  Interventions: Procedure: regional anesthesia
- regional anesthesia (Active Comparator)
  Interventions: Procedure: local anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — Regional anesthesia will be compared to local anesthesia
  Arms: Local anesthesia
Procedure: local anesthesia — Regional anesthesia will be compared to local anesthesia
  Arms: regional anesthesia

SUMMARY:
This study is being done to compare the two anesthesia techniques which are commonly used in the formation of arteriovenous fistulas: local anesthesia and regional anesthesia. Local anesthesia means that, your doctor will inject numbing medication directly into the tissue or part of your body where the surgery will be done. In this case, the numbing medication will be injected directly into the area where your fistula will be made. In regional anesthesia, the numbing medication will be injected around the nerve (part of the body that gives sensation) for your arm, to make the entire arm numb. The purpose of this study is to compare the three month success rates of AV fistulae created by the two anesthesia techniques.

DETAILED DESCRIPTION:
The primary objectives of the study are:

1. To evaluate the three-month success rate for AV fistulas constructed while using regional anesthesia against those constructed while using local anesthesia. Success will be evaluated by a dialysis access ultrasound, which will be performed three months after completion of the procedure. Successful will be defined as a mean blood flow of 600 ml/min and above, or receiving hemodialysis using the newly created AV fistula.
2. To evaluate the immediate (within 3 days) and long-term complications three months after AV fistula construction under regional anesthesia or local anesthesia.

The secondary objective of the study is to use a short questionnaire survey To assess patient comfort level after creation of AV fistula (e.g. nausea, analgesia).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years old
* Able to give informed consent
* Creation of first time AV fistula
* Possible 3 month follow up visit
* ASA-I-IV

Exclusion Criteria:

* BMI ≥40
* Repeated AV fistula creation,
* ASA -V,
* Allergic to local anesthetic agents,
* Significant lung and cardiac disease,
* Infection at the site of regional anesthesia,
* Pre-existing peripheral nerve damage,
* Significant bleeding disorders,

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
AV fistula success rate | Three months from the day of creation
  To evaluate the three-month success rate for AV fistulas constructed while using regional anesthesia against those constructed while using local anesthesia. Success will be evaluated by a dialysis access ultrasound, which will be performed three months after completion of the procedure. Successful will be defined as a mean blood flow of 600 ml/min and above, or receiving hemodialysis using the newly created AV fistula.

SECONDARY OUTCOMES:
Short term comfort level | Within three days of procedure
  To assess patient comfort level after creation of AV fistula (e.g. nausea, analgesia).
Short term safety, number of post operative complications | Three days after the creation
  b) To evaluate the immediate complications (within 3 days)after AV fistula construction under regional anesthesia or local anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States